CLINICAL TRIAL: NCT00763776
Title: Parenchyma Resection of Cirrhotic Liver by the Clamp Crushing Technique and the Ultrasonic Dissector : Randomized Comparative Study.
Brief Title: Parenchyma Resection of Cirrhotic Liver by the Clamp Crushing Technique and the Ultrasonic Dissector
Acronym: SECCI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty for the patient recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K070105
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2011-01

CONDITIONS: Liver Cirrhosis; Liver Neoplasms; Carcinoma, Hepatocellular
Keywords: Liver cirrhosis; Hepatectomy; Liver parenchyma transection; Randomized controlled trial
MeSH Terms: conditions — Liver Cirrhosis; Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Liver transection by clamp crushing technique
  Interventions: Device: clamp crushing technique
- 2 (Other): Liver transection by the ultrasonic dissector
  Interventions: Device: ultrasonic dissector

INTERVENTIONS:
Device: clamp crushing technique — Liver transection during hepatectomy by clamp crushing technique
  Arms: 1
Device: ultrasonic dissector — Liver transection during hepatectomy by the ultrasonic dissector
  Arms: 2

SUMMARY:
To identify the most efficient parenchyma transection technique for cirrhotic liver resection between the clamp crushing technique and the ultrasonic dissector.

Primary endpoint is intra-operative blood loss during liver transection (ml). Expected results and implications: If one of the technique is better than the other, surgical teams could prefer it to minimize the morbidity of liver resection in cirrhotic patients.

DETAILED DESCRIPTION:
Design Multicentric randomized controlled simple blinded trial comparing the clamp crushing technique vs. the ultrasonic dissector. The trial will last 24 months with 21 month-inclusion time.

Patients Patients will be enrolled in 5 university hospitals in Ile de France. Eligibility criteria include adults with Child A liver cirrhosis undergoing partial hepatectomy (≥ 1 liver segment). Exclusion criteria include non cirrhotic patients, Child B or C cirrhosis, portal hypertension and laparoscopic hepatectomy.

Sample size calculation was performed with the expectation of a 250 ml (one red cells pack) difference in blood loss during parenchyma transection with a level of statistical significance of 0.05 and a power of 0.80. These calculations indicated to include at least 60 patients in each group.

Secondary endpoints include blood loss standardized to the transection area (ml/cm²), free margins around the tumor, postoperative liver ischemia-reperfusion injury and postoperative complications.

Course of the study An informed consent will be obtained from each patient prior to surgery. Each patient will be randomized the day prior to surgery. As usual, each patient will be followed daily until he will discharge (10 days) and for 2 months at the postoperative outcome patient clinic, which will end the study period for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Child A liver cirrhosis
* Partial hepatectomy (≥ 1 segment).
* Patient at least 18 years of age

Exclusion Criteria:

* Non cirrhotic patient
* Child B or C cirrhosis
* Portal hypertension
* Laparoscopic hepatectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Intra-operative blood loss during liver transection (ml). | during liver transection

SECONDARY OUTCOMES:
Intra-operative blood loss standardized to the transection area (ml/cm²) | during liver transection
free margins around the tumor | during liver transection
postoperative liver ischemia-reperfusion injury (post-operative peak of transaminases) | daily until the discharge of the patient
60-day postoperative complications | 2 months after the liver transection

CONTACTS AND LOCATIONS:
Overall Officials: Mickael LESURTEL, MD-PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital BEAUJON, Clichy, France